CLINICAL TRIAL: NCT04659512
Title: Recurrent Neovascular Age-related Macular Degeneration After Discontinuation of VEGF Inhibitors Managed in a Treat and Extend Regimen
Brief Title: Recurrent Neovascular Age-related Macular Degeneration After Therapy Suspension
Status: Completed | Type: Observational
Sponsor: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Anders Kvanta, PI, St. Erik Eye Hospital
Other Study IDs: 20171
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate prospectively the recurrence rate of active macular neovascularization (MNV) and the visual outcome in patients with nAMD previously on a Treat and Extend regimen where treatment has been discontinued due to disease stability.

DETAILED DESCRIPTION:
All study subjects had nAMD and were treated at diagnosis with three monthly aflibercept injections and then subsequently followed in a treat and extend regimen with extensions by two weeks if no signs of disease activity were seen. Hemorrhage, intraretinal macular edema or subretinal fluid were considered signs of disease activity. Patients reaching 12-week intervals without any evidence of disease activity on three consecutive visits, a BCVA between 35-88 letters (Snellen 20/200- 20/20) and a near vision of at least 24 points were eligible for study inclusion.

If there were signs of recurrent disease activity during the follow-up, study participation was concluded at that point and intravitreal therapy was resumed. Between scheduled visits patients were encouraged to monitor their vision at home using monocular visual assessments and were advised to return earlier than planned if symptoms of visual deterioration or metamorphopsia occurred. At baseline and at every follow-up visit all patients had a full dilated ophthalmic examination. Optical coherence tomography (OCT) images were obtained by using the Zeiss Cirrus OCT instrument (Carl Zeiss Meditec, Inc.,Dublin, Ca). A pigment epithelial detachment (PED) was identified as an elevation of the RPE band and included both serous and fibrovascular PED. Near vision was tested at 40cm with the addition of +3 dioptres to the BCVA refraction. For near vision assessment we used the LIX adult A chart (Ortho-KM, Lund, Sweden) graded in typographical points, the largest text being 24 points and the smallest 4 points.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inactive neovascular AMD reaching 12-week intervals in a treat and extend regimen without any evidence of disease activity on three consecutive visits.
* BCVA between 35-88 letters (Snellen 20/200- 20/20)
* Near vision of at least 24 points

Exclusion Criteria:

• Active neovascular AMD

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inactive neovascular AMD reaching 12-week intervals in a treat and extend regimen without any evidence of disease activity on three consecutive visits.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-06-06 (Actual)

PRIMARY OUTCOMES:
Disease recurrence | 12 months
  The proportion of patients with recurrent disease within 12 months after the last injection.

SECONDARY OUTCOMES:
Risk factors for disease recurrence | 12 months
  Effect of age, lesion type, anatomic parameters (PED, geographic atrophy (GA) and sub macular fibrosis), previous episodes of recurrence and total number of injections before suspension, on risk of reactivation.
Visual outcome | 12 months
  Change in BCVA at time of recurrence and after resumed therapy.

CONTACTS AND LOCATIONS:
Overall Officials: David Epstein, Principal Investigator — Sankt Erik Eye Hospital
Locations (1):
- St Eriks Eye Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No